CLINICAL TRIAL: NCT02726997
Title: Matched Paired Pharmacodynamics and Feasibility Study of Durvalumab in Combination With Chemotherapy in Frontline Ovarian Cancer (N-Dur)
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-0900; NCI-2016-00557 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2015-0900 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2016-03-24; First posted 2016-04-04 (Estimated); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Stage III Fallopian Tube Cancer AJCC v7; Stage III Ovarian Cancer AJCC v6 and v7; Stage III Primary Peritoneal Cancer AJCC v7; Stage IIIA Fallopian Tube Cancer AJCC v7; Stage IIIA Ovarian Cancer AJCC v6 and v7; Stage IIIA Primary Peritoneal Cancer AJCC v7; Stage IIIB Fallopian Tube Cancer AJCC v7; Stage IIIB Ovarian Cancer AJCC v6 and v7; Stage IIIB Primary Peritoneal Cancer AJCC v7; Stage IIIC Fallopian Tube Cancer AJCC v7; Stage IIIC Ovarian Cancer AJCC v6 and v7; Stage IIIC Primary Peritoneal Cancer AJCC v7; Stage IV Fallopian Tube Cancer AJCC v6 and v7; Stage IV Ovarian Cancer AJCC v6 and v7; Stage IV Primary Peritoneal Cancer AJCC v7
MeSH Terms: conditions — Fallopian Tube Neoplasms | interventions — Carboplatin; durvalumab; Immunoglobulin G; Disulfides; Paclitaxel; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (durvalumab, carboplatin, paclitaxel, questionnaire) (Experimental): NEOADJUVANT CHEMOTHERAPY: Before debulking surgery, patients receive durvalumab and carboplatin IV over 1 hour on day 1, and paclitaxel IV over 3 hours on days 1, 8, and 15. Treatment repeats every 21 days for up to 3 courses in the absence of disease progression or unacceptable toxicity. Patients then undergo debulking surgery.
  SURGERY: After 3 courses of chemotherapy, patients undergo debulking laparoscopic surgery.
  ADJUVANT THERAPY: Beginning after debulking surgery, patients receive carboplatin IV over 1 hour on day 1, paclitaxel IV over 3 hours on days 1, 8, and 15, and durvalumab IV over 1 hour on day 1. Treatment repeats every 21 days for up to 3 courses in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE THERAPY: Patients receive durvalumab IV over 1 hour on day 1 and 15. Treatment repeats every 28 days for up to 7 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Carboplatin; Biological: Durvalumab; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel; Other: Pharmacological Study; Other: Quality-of-Life Assessment

INTERVENTIONS:
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Biological: Durvalumab — Given IV
  Other Names: Imfinzi; Immunoglobulin G1, Anti-(Human Protein B7-H1) (Human Monoclonal MEDI4736 Heavy Chain), Disulfide with Human Monoclonal MEDI4736 Kappa-chain, Dimer; MEDI-4736; MEDI4736
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Other: Pharmacological Study — Correlative studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This phase I/II trial studies how well durvalumab works when given in combination with carboplatin and paclitaxel in treating patients with stage III-IV ovarian, primary peritoneal, or fallopian tube cancer. Immunotherapy with monoclonal antibodies, such as durvalumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Drugs used in chemotherapy, such as carboplatin and paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving durvalumab in combination with carboplatin and paclitaxel may be a better treatment for ovarian, primary peritoneal, or fallopian tube cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To explore basal levels and effects of durvalumab in combination with chemotherapy on molecular markers in immune-related pathways, including but not limited to, deoxyribonucleic acid (DNA) copy number, mutation, and level of ribonucleic acid (RNA) and protein expression, before and after durvalumab and chemotherapy treatment in women with primary advanced high grade serous ovarian, fallopian tube, or primary peritoneal cancer.

SECONDARY OBJECTIVES:

I. To evaluate progression-free survival of paclitaxel and carboplatin and durvalumab in patients with advanced stage, metastatic ovarian cancer undergoing neoadjuvant chemotherapy.

II. To describe the feasibility of combination therapy and maintenance durvalumab in this population.

III. To evaluate the safety, tolerability and pharmacokinetics (PK) of combination and maintenance durvalumab.

IV. To report overall survival.

EXPLORATORY OBJECTIVES:

I. To evaluate circulating lymphoid populations (subsets). II. To determine tissue programmed death-ligand 1 (PD-L1) expression and T-cell infiltration.

III. To measure circulating immune-related cytokines/chemokines. IV. To capture patient reported outcomes (symptoms, quality of life, and patient utilities).

OUTLINE:

NEOADJUVANT CHEMOTHERAPY: Before debulking surgery, patients receive durvalumab and carboplatin intravenously (IV) over 1 hour on day 1, and paclitaxel IV over 3 hours on days 1, 8, and 15. Treatment repeats every 21 days for up to 3 courses in the absence of disease progression or unacceptable toxicity. Patients then undergo debulking surgery.

SURGERY: After 3 courses of chemotherapy, patients undergo debulking laparoscopic surgery.

ADJUVANT THERAPY: Beginning after debulking surgery, patients receive carboplatin IV over 1 hour on day 1, paclitaxel IV over 3 hours on days 1, 8, and 15, and durvalumab IV over 1 hour on day 1. Treatment repeats every 21 days for up to 3 courses in the absence of disease progression or unacceptable toxicity.

MAINTENANCE THERAPY: Patients receive durvalumab IV over 1 hour on day 1 and 15. Treatment repeats every 28 days for up to 7 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days, 2, 3, 4, 6, 8, 9, 10, and 12 months, and then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent and any locally-required authorization (e.g., Health Information Portability and Accountability Act [HIPAA] in the United States of America [USA], European Union [EU] Data Privacy Directive in the EU) obtained from the subject prior to performing any protocol-related procedures, including screening evaluations
* Histology showing high-grade epithelial non-mucinous ovarian, primary peritoneal, or fallopian tube cancer
* No prior treatment for primary advanced (stage III or IV) epithelial ovarian, primary peritoneal, or fallopian tube carcinoma such as irradiation, chemotherapy, hormonal therapy, immunotherapy, investigational therapy, surgery, and/or other concurrent agents or therapies
* A disposition to neoadjuvant chemotherapy with planned interval tumor reductive surgery after 3 complete cycles of treatment
* Planned chemotherapy with combination carboplatin and paclitaxel given intravenously
* Have measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1

  * Measurable disease is defined at least one lesion that can be accurately measured in at least one dimension (longest dimension to be recorded); each target lesion must be > 20 mm when measured by conventional techniques, including palpation, plain x-ray, computed tomography (CT), and magnetic resonance imaging (MRI), or > 10 mm when measured by spiral CT
  * Patients with non-measurable but evaluable solid tumors may be deemed eligible contingent upon principal investigator (PI) review; a non-measurable but evaluable solid tumor is defined as either unidimensionally measurable lesions, masses with margins not clearly defined, or lesions with maximal perpendicular diameters < 10 mm that can still be evaluated for the primary endpoint
* Peripheral neuropathy grade 0 or 1 by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.03
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Life expectancy >= 12 weeks
* Hemoglobin (Hgb) >= 9 g/dL
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L (> 1500 per mm^3)
* Platelet count >= 100 x 10^9/L (> 100,000 per mm^3)
* Serum bilirubin =< 1.5 x institutional upper limit of normal (ULN)
* Aspartate Transaminase (AST) and alanine transaminase (ALT) =< 2.5 x institutional upper limit of normal (ULN) unless liver metastases are present, in which case it must be =< 5 x ULN
* Serum creatinine clearance (CL) > 40 mL/min by the Cockcroft-Gault formula or by 24-hour urine collection for determination of creatinine
* Subjects must either be of non-reproductive potential (i.e., post-menopausal by history: >= 60 years old and no menses for >= 1 year without an alternative medical cause; OR history of hysterectomy, OR history of bilateral tubal ligation, OR history of bilateral oophorectomy) or must have a negative serum pregnancy test upon study entry
* Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up
* Pre-treatment tumor tissue available for research purposes; this tissue can be collected from preoperative laparoscopy, other diagnostic biopsy, or a research-specific biopsy; this pre-treatment tumor must be amenable to repeat tissue sampling after induction therapy
* Signed informed consent on protocol LAB02-188
* For participation in the patient-reported outcomes and qualitative interviews, subjects must be fluent in English

Exclusion Criteria:

* Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site)
* Previous enrollment in the present study
* Prior treatment for ovarian, fallopian tube, or primary peritoneal cancer
* Histology showing mucinous or low grade epithelial carcinoma
* Participation in another clinical study with an investigational product during the last 4 weeks
* Any previous treatment with a programmed cell death protein 1 (PD1) or programmed cell death ligand 1 (PD-L1) inhibitor, including durvalumab
* History of another primary malignancy except for: malignancy treated with curative intent and with no known active disease >= 5 years before the first dose of study drug and of low potential risk for recurrence; adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease; or adequately treated carcinoma in situ without evidence of disease e.g., cervical cancer in situ
* Mean QT interval corrected for heart rate (QTc) >= 470 ms calculated from 3 electrocardiograms (ECGs) using Bazett's correction
* Current or prior use of immunosuppressive medication within 28 days before the first dose of durvalumab, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid
* Any unresolved toxicity (> CTCAE grade 2) from previous anti-cancer therapy; any prior grade >= 3 immune-related adverse event (irAE) while receiving any previous immunotherapy agent, or any unresolved irAE > grade 1
* Active or prior documented autoimmune disease within the past 2 years; NOTE: Subjects with vitiligo, Grave's disease, or psoriasis not requiring systemic treatment (within the past 2 years) are not excluded
* Active or prior documented inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis)
* History of primary immunodeficiency
* History of allogeneic organ transplant
* History of hypersensitivity to durvalumab or any excipient
* History of hypersensitivity to paclitaxel or carboplatin or their excipients
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease or gastritis, active bleeding diatheses including any subject known to have evidence of acute or chronic hepatitis B, hepatitis C or human immunodeficiency virus (HIV), or psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the subject to give written informed consent
* Known history of previous clinical diagnosis of tuberculosis
* History of leptomeningeal carcinomatosis
* Receipt of live attenuated vaccination within 30 days prior to study entry or within 30 days of receiving durvalumab
* Female subjects who are pregnant/breast-feeding or who are of reproductive potential and not employing acceptable methods of birth control; acceptable methods of contraception include true abstinence in line with the preferred and usual lifestyle choice of the patient, tubal ligation, vasectomized partner, barrier methods (e.g., cap plus spermicide, sponge plus spermicide, diaphragm plus spermicide, or male condom plus a spermicide), intrauterine device methods (e.g., Copper T or Levonorgestrel-releasing intrauterine system), or hormonal methods (e.g., any registered and marketed contraceptive agent that contains an estrogen and/or a progestational agent) and that is administered via the oral, subcutaneous, transdermal, intrauterine, or intramuscular route as an implant, hormone shot or injection, combined pill, minipill or patch; all methods of contraception should be used in combination with the use of a condom by their male sexual partner for intercourse
* Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results
* Symptomatic or uncontrolled brain metastases requiring concurrent treatment, inclusive of but not limited to surgery, radiation and/or corticosteroids
* Subjects with uncontrolled seizures

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-07-06 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Pharmacodynamic Changes Induced by Treatment with Durvalumab in Combination with Paclitaxel and Carboplatin in Women with Advanced Stage, Metastatic Ovarian Cancer Using Paired T-Test | 1 year
  Paired t-test with a 2-sided significance level of 0.05 used to test whether the change in biomarker expression from pre-treatment to post-treatment with Durvalumab is different from 0.
Pharmacodynamic Changes Induced by Treatment with Durvalumab in Combination with Paclitaxel and Carboplatin in Women with Advanced Stage, Metastatic Ovarian Cancer Using an Exact Binomial Test | 1 year
  Exact binomial test with a 1-sided significance level of 0.05 used to test whether the probability of a biomarker increasing (or decreasing) is > 0.50.
Pharmacodynamic Changes Induced by Treatment with Durvalumab in Combination with Paclitaxel and Carboplatin in Women with Advanced Stage, Metastatic Ovarian Cancer | 1 year
  Fisher's exact test with a 1-sided significance level of 0.05 used to compare the proportion of participants treated with Durvalumab who have increasing (or decreasing) expression rates with the corresponding proportion from a historical control group of 30 untreated patients.
Pharmacodynamic Changes Induced by Treatment with Durvalumab in Combination with Paclitaxel and Carboplatin in Women with Advanced Stage, Metastatic Ovarian Cancer Using a 2-Sample T-Test | 1 year
  A 2-sample t-test with a 2-sided significance level of 0.05 used to compare change in biomarker expression between patients treated with Durvalumab and a control group of 30 untreated patients.

SECONDARY OUTCOMES:
Progression-Free Survival with Treatment with Durvalumab in Combination with Paclitaxel and Carboplatin in Women with Advanced Stage, Metastatic Ovarian Cancer | 1 year
  Progression defined by any of the following: 25% increase in sum of the products of perpendicular diameters of enhancing lesions compared with the smallest tumor measurement obtained either at baseline (if no decrease) or best response, on stable or increasing doses of corticosteroids; significant increase in T2/FLAIR nonenhancing lesion on stable or increasing doses of corticosteroids compared with baseline scan or best response after initiation of therapy not caused by comorbid events (eg, radiation therapy, demyelination, ischemic injury, infection, seizures, postoperative changes, or other treatment effects); any new lesion; clear clinical deterioration not attributable to other causes apart from the tumor (eg, seizures, medication adverse events, complications of therapy, cerebrovascular events, infection) or changes in corticosteroid dose; failure to return for evaluation as a result of death or deteriorating condition; or clear progression of nonmeasurable disease.
Feasibility of Treatment with Durvalumab in Combination with Paclitaxel and Carboplatin in Women with Advanced Stage, Metastatic Ovarian Cancer Determined by Methods of Thall et all | 126 days
  Feasibility defined as the ability to complete all planned cycles of adjuvant therapy, using the methods of Thall et al. (1994).

CONTACTS AND LOCATIONS:
Overall Officials: Shannon N Westin, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org